CLINICAL TRIAL: NCT00665990
Title: Phase I Study of Bevacizumab and Sorafenib Combined With Low Dose Cyclophosphamide in Patients With Refractory Solid Tumors and Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANGIO1; NCI-2011-01146 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Refractory Solid Tumors; Leukemia
MeSH Terms: conditions — Leukemia | interventions — Bevacizumab; Sorafenib; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): All participants will receive bevacizumab, sorafenib, and cyclophosphamide until maximum tolerated dose is reached.
  Interventions: Drug: Bevacizumab; Drug: Sorafenib; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab starting dose of 5 mg/kg every 3 weeks increasing in combination with Sorafenib and Cyclophosphamide until maximum tolerated dose
  Other Names: rhuMab VEGF; Avastin(R)
Drug: Sorafenib — Sorafenib 90 mg/m2 PO every 12 hours increasing in combination with Bevacizumab and Cyclophosphamide until maximum tolerated dose
  Other Names: BAY-43-9006; Nexavar(R)
Drug: Cyclophosphamide — Cyclophosphamide 50 mg/m2 PO once daily increasing in combination with Bevacizumab and Sorafenib until maximum tolerated dose
  Other Names: Cytoxan(R)

SUMMARY:
Phase I Study of Bevacizumab and Sorafenib Combined with Low Dose Cyclophosphamide in Patients with Refractory Solid Tumors and Leukemia. Patients with solid tumors (including central nervous tumors) that are recurrent or refractory to standard therapy, or for whom standard therapy is not available. Once a maximum tolerated dose (MTD) has been established in patients with recurrent or refractory solid tumors, the tolerability of this dose will be tested in patients with refractory or recurrent leukemia and an expanded cohort of patients with refractory or recurrent solid tumors.

DETAILED DESCRIPTION:
Phase I Study of Bevacizumab and Sorafenib Combined with Low Dose Cyclophosphamide in Patients with Refractory Solid Tumors and Leukemia. Patients with solid tumors (including central nervous tumors) that are recurrent or refractory to standard therapy, or for whom standard therapy is not available. Once a maximum tolerated dose (MTD) has been established in patients with recurrent or refractory solid tumors, the tolerability of this dose will be tested in a maximum of 6 patients, in cohorts of 3, with refractory or recurrent leukemia and a maximum of 24 evaluable patients, in cohorts of 6, with refractory or recurrent solid tumors.

Approximately 21-24 patients with refractory solid tumors to define the maximum tolerated dose (MTD) and 6 patients with recurrent or refractory leukemia,12 patients with refractory or recurrent bone or soft tissue sarcomas and 12 patients with other refractory or recurrent solid tumors (including lymphomas) to test the tolerability of this MTD in patients with hematological malignancies. Bevacizumab will be administered intravenously at a starting dose of 5 mg/kg every 3 weeks with sorafenib by mouth every 12 hrs at a starting dose of 90 mg/m2 every 12 hours and cyclophosphamide by mouth daily at a dose of 50 mg/m2/day (dose level 1). A course of therapy will be considered to be of 21 days duration. Once a maximum tolerated dose of sorafenib (sMTD) in combination with bevacizumab and cyclophosphamide has been determined, 6 patients with recurrent or refractory leukemia will be then be evaluated at the solid tumor MTD to test the tolerability of this combination in patients with hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

NOTE: As of May 2013, enrollment of solid tumor participants was completed. Participants with a diagnosis of leukemia continue to be enrolled.

* Diagnosis: Solid tumors, including central nervous system tumors and lymphomas, that are recurrent or refractory to standard therapy or for which there is no standard therapy. Histologic verification of diagnosis is required.
* Age: < or = 21 years of age at the time of original diagnosis
* Life expectancy: at least 8 weeks
* Performance status: Karnofsky > or = 50 for > 10 years of age; Lansky > or = 50 for children < or = 10 years of age.
* Organ Function: Must have adequate organ and marrow function
* Prior Therapy: Patient must have fully recovered from the acute toxic effects of all prior therapy prior to enrolling on study.
* Must not have current or recent use of full-dose anticoagulants
* Must not have received medications known to inhibit platelet function or known to selectively inhibit cyclooxygenase-2 (COX-2) activity
* Bevacizumab and sorafenib should not be administered to pregnant women.
* Pregnancy tests must be obtained in girls who are > 10 years of age or post-menarchal.
* Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Breast feeding should be discontinued if a mother wishes to participate in this study.
* Patients with a documented, chronic non-healing wound, ulcer, or bone fracture or history of a major surgical procedure or significant traumatic injury within 28 days prior to beginning therapy should be excluded due to preclinical evidence supporting the potential for delayed wound healing.
* Patients must not have a deep venous or arterial thrombosis (including pulmonary embolism) within the last three months prior to study entry, and must not have a known thrombophilic condition
* Patients must not have a history of myocardial infarction, severe or unstable angina, or severe peripheral vascular disease.
* Ability to understand and willingness of research participant or legal guardian/representative to give written informed consent.

Exclusion Criteria:

* Body surface area < 0.3 m2
* Presence of a known bleeding diathesis or coagulopathy
* Patients with evidence of intra-tumoral central nervous system hemorrhage. in current scans. Patients are required to have a head CT or MRI within 2 weeks prior to study enrollment.
* Patients with known hypersensitivity to other recombinant human antibodies
* Patients who have an uncontrolled infection
* Patients with recurrent or refractory leukemia will be excluded from the dose escalation component of the phase I trial.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2007-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose and dose limiting toxicity of bevacizumab and sorafenib administered in combination with low dose cyclophosphamide to patients with refractory solid tumors. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sara Federico, MD, Principal Investigator — St. Jude Children' Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] McCarville MB, Coleman JL, Guo J, Li Y, Li X, Honnoll PJ, Davidoff AM, Navid F. Use of Quantitative Dynamic Contrast-Enhanced Ultrasound to Assess Response to Antiangiogenic Therapy in Children and Adolescents With Solid Malignancies: A Pilot Study. AJR Am J Roentgenol. 2016 May;206(5):933-9. doi: 10.2214/AJR.15.15789. Epub 2016 Mar 21. PMID 26999488
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols